CLINICAL TRIAL: NCT02212886
Title: A Prospective 1-year, Open-label, Two Arms, Multicenter, Phase IIa Study to Assess Safety, Tolerability and Efficacy of Once a Month Long-acting Intramuscular Injection of 80 or 40 mg Glatiramer Acetate (GA Depot) in Subjects With Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: Safety, Tolerability and Efficacy of Monthly Long-acting IM Injection of 80 or 40 mg GA Depot in Subjects With RRMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mapi Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI GA Depot - 001
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Glatiramer acetate; Copaxone®; Multiple sclerosis; Relapsing remitting multiple sclerosis; RRMS; GA Depot; Monthly injection
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GA Depot 80mg (Experimental): Monthly IM injection
  Interventions: Drug: GA Depot 80 mg
- GA Depot 40mg (Experimental): Monthly IM injection
  Interventions: Drug: GA Depot 40 mg

INTERVENTIONS:
Drug: GA Depot 80 mg — Recruitment completed
  Other Names: Microspheres containing GA
  Arms: GA Depot 80mg
Drug: GA Depot 40 mg — Recruitment completed
  Other Names: Microspheres containing GA
  Arms: GA Depot 40mg

SUMMARY:
* This is a phase IIa study in which GA Depot 80 or 40mg is administered as an IM injection to subjects with RRMS at 4 week intervals for 52 weeks of treatment.
* The purpose of the study is to assess safety, tolerability, and efficacy of a monthly long-acting IM injection of 80 or 40mg GA Depot in subjects with RRMS. The study will include subjects switching from daily or thrice weekly administration of 20 mg or 40mg respectively of glatiramer acetate (GA, i.e., Copaxone®) injection

DETAILED DESCRIPTION:
* 25 Subjects with a diagnosis of relapsing remitting multiple sclerosis (RRMS) who are treated with daily or thrice weekly subcutaneous injections of 20 mg or 40 mg respectively of GA (Copaxone®) during the previous 12 months
* Study product is GA long-acting injection (GA Depot) which is a combination of extended-release microspheres for injection and diluent (water for injection) for parenteral use. GA Depot will be administered intramuscularly (IM).
* The study duration for an individual subject in the core study will be 60 weeks, consisting of 4 weeks of screening evaluation (weeks -4 to 0), followed by a 52-week open-label treatment period, and a 4 weeks follow up period: through a total of 17 visits.
* For both arms, subjects who completed 13 injections and who consented (by signing an informed consent) are able to enter the optional 8 years extension period. During the extension period subjects will receive 40 mg of GA Depot IM once every 4 weeks.
* Physical, vital signs and safety assessment - will be performed at each visit during the whole study. Physical examination will be performed quarterly during the extension period.
* MRI at visit 1 (screenings), at week 24, week 52 (end of core study) and every 6 months during the extension period.
* Neurological and safety laboratory tests at screening visit, on visits in weeks 4, 12, 24, 36, 52 (end of core study) and every 6 months during the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a diagnosis of RRMS.
* Diagnosis of multiple sclerosis (MS) consistent with the McDonald Criteria (revisions of 2010).
* Treatment with 20 mg or 40 mg of GA (Copaxone®) during the previous 12 months with ongoing treatment at the Screening Visit.
* Normal renal function.
* Normal liver function.
* Normal hemoglobin concentration.
* Absence of any clinically significant medical, psychiatric or laboratory abnormalities.
* Ability to provide written informed consent.

Exclusion Criteria:

* Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the investigator, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
* Concomitant Autoimmune disease.
* Severe anemia (hemoglobin < 10 g/dL).
* Abnormal renal function (serum creatinine > 1.5xULN).
* Abnormal liver function (transaminases >2xULN).
* Pregnant or breast-feeding women.
* Women capable of child bearing must have a negative urine pregnancy test at screening visit and use an adequate contraceptive method throughout the study. Women who are surgically sterile (hysterectomy or tubal ligation) or whose last menstruation was 12 months or more prior to the Screening Visit are considered to be of non-child-bearing potential. Acceptable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; estrogen patch; and adequate barrier methods in conjunction with spermicide. Abstinence is considered an acceptable contraceptive regimen.
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study drug, e.g. GA, polylactic-co-glycolic acid (PLGA), polyvinyl alcohol (PVA).
* Known or suspected history of drug or alcohol abuse.
* Positive test for HIV, hepatitis, venereal disease research laboratory test (VDRL), or tuberculosis.
* Participation in an investigational drug study within 30 days prior to start of this study.
* Active malignant disease of any kind. However, a patient, who has had a malignant disease in the past, was treated and is currently disease - free for at least 5 years, may be considered to be enrolled in the study. In this case the sponsor medical expert approval is required.
* Treatment with any kind of steroids during the last 30 days.
* Confirmed relapse during the last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Safety / Adverse events | During the study (1 year treatment)
  Number of patients experiencing adverse events and assessments of localized skin reactions at injection sites.

SECONDARY OUTCOMES:
Efficacy/Change in Relapse Rate | During the study (1 year treatment)
  Relapse rate detected during the study compared to relapse rate observed in the 12 months prior to study start.
Efficacy/Changes in brain MRI | During the study (1 year treatment)
  Changes from baseline to end of treatment visit in the number of enhancing lesions and new lesions images of brain MRI
Efficacy/Changes in EDSS | 1 year
  Change from baseline to end of treatment visit of Expanded Disability Status Scale (EDSS) score.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Flechter, M.D, Principal Investigator
Locations (3):
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - TASMC, Tel Aviv